CLINICAL TRIAL: NCT04480749
Title: Syphilis Self-testing to Expand Test Uptake Among Men Who Have Sex With Men (SST)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Biomedical Research and Training Institute, Zimbabwe (Other); Pangaea Zimbabwe Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17848
Record Dates: First submitted 2020-07-02; First posted 2020-07-21 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-03

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Testing (Other): Among men in the control group, they will receive a list of local clinics that can provide free syphilis testing.
  Interventions: Diagnostic Test: Access to Facility based Syphilis Testing
- Self-Testing (Experimental): In the intervention arm we will provide a treponemal rapid syphilis test kit to all individuals in the intervention arm of the pilot, delivered through MSM community facilitators. This is similar to existing rapid treponemal test kits that are available at many clinical facilities. Kits will be accompanied by simplified pictorial instructions on finger prick blood sample collection.
  Interventions: Diagnostic Test: Access to Facility based Syphilis Testing; Diagnostic Test: Syphilis Self-Test

INTERVENTIONS:
Diagnostic Test: Access to Facility based Syphilis Testing — List of facilities where syphilis testing can be accessed
Diagnostic Test: Syphilis Self-Test — Rapid Treponemal Test kit
  Arms: Self-Testing

SUMMARY:
Syphilis infection is a major global health problem, leading to substantial morbidity among key populations in low- and middle-income countries (LMICs). Men who have sex with men (MSM) are disproportionately affected by syphilis worldwide. Rates of syphilis diagnoses have been increasing amongst MSM in many countries in the last decade. A growing evidence base supporting HIV self-testing shows that self-testing kits based on the same proposed clinical pathways are feasible and reliable. The proposed study will leverage this body of evidence and apply it to syphilis self-testing.

This is a pilot study conducted in Zimbabwe. It aims to collect initial data on the feasability of implementing syphilis self-testing to establish if a large scale-RCT of this approach would be appropriate and, if so, to inform the design of this trial.

The investigators will recruit 100 MSM in Harare to join the pilot program. Participants will be recruited through two methods: in-person at MSM community-based organizations that currently operate HIV self-testing programs and online through banner advertisements that advertise HIV self-testing.

Study Arms:

Arm 1: One arm of the pilot will receive a free syphilis self-test kit (Intervention Arm) Arm 2: One arm will receive standard free facility-based syphilis testing (Control Arm).

Intervention:

In the intervention arm the investigators will provide a treponemal rapid syphilis test kit to all participants in the intervention arm of the pilot, delivered through MSM community facilitators. This is similar to existing rapid treponemal test kits that are available at many clinical facilities. Kits will be accompanied by simplified pictorial instructions on finger prick blood sample collection. Among participants in the control group, they will receive a list of local clinics that can provide free syphilis testing.

Data Collection:

For individuals in the intervention am the investigators will aim to obtain confirmation of test uptake. This will be done using either photographic confirmation sent via encrypted message on a smartphone, SMS message of a unique code or sending a unique five-digit code along with their test result to the study coordinator. The investigators will conduct cross-sectional surveys at baseline and six months later to assess sexual risk behaviours, HIV and syphilis testing experiences, and self-testing experiences. In addition to the survey data tool the investigators will conduct in-depth interviews with a small number of participants to gain additional data about their experience of syphilis self-testing.

The investigators will obtain information on linkage to care from routine clinic administrative records and by providing study participants with a unique code to be provided when attending at the facility.

Analysis:

The investigators will used mixed-methods to evaluate our pilot intervention including

The investigators will examine the proportion of individuals who undertake a syphilis test in the interventional and control arms; among those who receive a test, the proportion of individuals who receive appropriate post-testing services. The investigators will also collect qualitative data on attitudes to syphilis self-testing and quantitative data on syphilis prevalence to inform a subsequent clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men
* Able to consent

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with men
Enrollment: 100 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harare City Council Health Facilities, Harare, NIL Return, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Routine Testing | Self-Testing
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Testing | Self-Testing | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 50 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Zimbabwe | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Syphilis Tests Undertaken
Description: The total number of participants undertaking a syphilis test
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Testing | Self-Testing
Number analyzed (Participants) | 50 | 50
Participants | 29 | 37

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Routine Testing | Self-Testing
All-Cause Mortality (participants affected / at risk) | 0/50 | 9/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT04480749/Prot_SAP_000.pdf